CLINICAL TRIAL: NCT00374907
Title: Mechanism of Action and Efficacy of Saxagliptin (BMS-477118) in the Treatment of Type 2 Diabetic Patients
Brief Title: A Study Assessing Saxagliptin Treatment in Subjects With Type 2 Diabetes Who Are Not Controlled With Diet and Exercise
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV181-041
Record Dates: First submitted 2006-09-07; First posted 2006-09-12 (Estimated); Results first posted 2011-01-21 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Saxagliptin (A) (Experimental): Metformin 500-1500 mg (open-label, as needed for rescue in LT)
  Interventions: Drug: Saxagliptin
- Placebo (ST) / Metformin (LT) (B) (Placebo Comparator): Metformin 500-1500 mg (open-label, as needed for rescue in LT)
  Interventions: Drug: Placebo; Drug: Metformin (blinded); Drug: Metformin (open-label)

INTERVENTIONS:
Drug: Saxagliptin — Tablet, Oral, 5 mg, Once daily, (up to 12 weeks ST, up to 104 weeks LT)
  Other Names: BMS-477118
  Arms: Saxagliptin (A)
Drug: Placebo — Tablet, Oral, 0 mg, Once daily (up to 12 weeks ST)
  Arms: Placebo (ST) / Metformin (LT) (B)
Drug: Metformin (blinded) — Tablet, Oral, 500 mg titrated to 1000 mg, Once daily (up to 104 weeks LT, starting at Week 12)
  Arms: Placebo (ST) / Metformin (LT) (B)
Drug: Metformin (open-label) — Tablets, Oral, 500-1500 mg, as needed (starting in LT)
  Arms: Placebo (ST) / Metformin (LT) (B)

SUMMARY:
The purpose of this clinical research study is to learn whether Saxagliptin can improve the body's ability to make its own insulin and lower blood sugar in people with type 2 diabetes

DETAILED DESCRIPTION:
All subjects will participate in a lead-in period, and qualifying subjects will continue into a short-term randomized treatment period. Subjects who complete the short-term period will be eligible to enter the long term extension period. Also, subjects who have an elevated blood sugar that requires additional medication for blood sugar control will be eligible to receive open-label metformin added onto their blinded study medication

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Drug naive
* Hemoglobin A1c (HbA1c) ≥6.0% and ≤8.0%
* Fasting C-peptide ≥1.0 ng/mL
* Body mass index ≤40 kg/m²

Exclusion Criteria:

* Recent cardiac or cerebrovascular event
* Elevated serum creatinine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2006-09; Primary Completion 2008-01 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Va San Diego Healthcare System, San Diego, California
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Diabetes & Glandular Disease Research Assoc,, Inc., San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 156 participants were enrolled in the study; 110 participants failed screening; 10 subjects entered lead-in and discontinued prior to randomization.
Groups:
- Saxagliptin 5 mg: Tablet, Oral, 5 mg, once daily, up to 12 weeks (short-term) and up to 104 weeks (long-term). Metformin 500-1500 mg (open-label, as needed for rescue in LT).
- Placebo / Metformin: Placebo Tablet, Oral, 0 mg, once daily, up to 12 weeks; Metformin Tablet, Oral, 500 mg/1000 mg, once daily, up to 104 weeks starting at Week 12 (end of ST period). Metformin 500-1500 mg (open-label, as needed for rescue in LT).
Period: 12-Week Short-term Period
Arm/Group | Saxagliptin 5 mg | Placebo / Metformin
Started | 20 | 16
Completed | 17 | 15
Not Completed | 3 | 1
Not completed — Subject Withdrew Consent | 3 | 1
Period: 116-Week Short-term + Long-term Period
Arm/Group | Saxagliptin 5 mg | Placebo / Metformin
Started | 20 | 16
Completed 12-week Short Term Period | 17 | 15
Completed | 7 | 2
Not Completed | 13 | 14
Not completed — Subject Withdrew Consent | 8 | 9
Not completed — Lack of Efficacy | 4 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Saxagliptin 5 mg: Tablet, Oral, 5 mg, once daily, up to 12 weeks (short-term) and up to 104 weeks (long-term)
- Placebo / Metformin: Placebo Tablet, Oral, 0 mg, once daily, up to 12 weeks; Metformin Tablet, Oral, 500 mg/1000 mg, once daily, starting at Week 12 and up to 104 weeks
- Total: Total of all reporting groups
Arm/Group | Saxagliptin 5 mg | Placebo / Metformin | Total
Number analyzed (Participants) | 20 | 16 | 36
Age, Continuous [Median (Full Range); unit: years] | 58 [43 to 69] | 55 [45 to 69] | 55.5 [43 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 8 | 6 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  White | 16 | 12 | 28
  Black/African American | 3 | 4 | 7
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  North America | 20 | 16 | 36
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 33.36 [24.67 to 39.35] | 32.31 [25.56 to 38.55] | 33.01 [24.67 to 39.35]

OUTCOME MEASURES:

1. Primary Outcome: Insulin Secretion Rate Area Under the Curve (AUC) During Intravenous (IV)-Oral Hyperglycemic Clamp - Percent Change From Baseline at Week 12
Description: Adjusted percent change in the insulin secretion rate AUC during a hyperglycemic clamp with an enteral glucose load [intravenous-oral hyperglycemic clamp (180-480 minutes)] at Week 12. The method used for calculating the insulin secretion rate was C-peptide deconvolution.
Time Frame: Baseline, Week 12
Population: Randomized participants with both a baseline and post-baseline value (up to Week 12).
Measure: Geometric Mean (95% Confidence Interval); unit: Percent Change (Percentage of Baseline)
Groups:
- Short Term Period: Saxagliptin 5 mg: Tablet, Oral, 5 mg, once daily, up to 12 weeks
- Short Term Period: Placebo: Tablet, Oral, 0 mg, once daily, up to 12 weeks
Arm/Group | Short Term Period: Saxagliptin 5 mg | Short Term Period: Placebo
Number analyzed (Participants) | 16 | 15
Percent Change (Percentage of Baseline) | 15.9 [4.2 to 29.0] | -2.2 [-12.4 to 9.3]
Statistical Analysis 1: Comparison: Short Term Period: Saxagliptin 5 mg vs Short Term Period: Placebo; Test type: Superiority or Other; p = 0.0350, ANCOVA — Between-group comparisons significant at alpha = 0.05, significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted percent difference for saxagliptin 5 mg vs placebo in Week 12 (LOCF) to baseline ratio. Adjusted for baseline; Adjusted Percent Difference = 18.5, 95% CI 2-sided [1.3 to 38.7] — ANCOVA model: logarithm(post/pre) = logarithm(pre) treatment

2. Secondary Outcome: Insulin Secretion Rate AUC During IV Hyperglycemic Clamp - Percent Change From Baseline at Week 12
Description: Adjusted percent change in the insulin secretion rate AUC during an intravenous hyperglycemic clamp (120-180 minutes) at Week 12. The method used for calculating the insulin secretion rate was C-peptide deconvolution.
Time Frame: Baseline, Week 12
Population: Randomized Participants with both a baseline and post-baseline value (up to Week 12).
Measure: Geometric Mean (95% Confidence Interval); unit: Percent Change (Percentage of Baseline)
Arm/Group | Short Term Period: Saxagliptin 5 mg | Short Term Period: Placebo
Number analyzed (Participants) | 18 | 16
Percent Change (Percentage of Baseline) | 22.6 [7.2 to 40.4] | -4.1 [-17.4 to 11.2]
Statistical Analysis 1: Comparison: Short Term Period: Saxagliptin 5 mg vs Short Term Period: Placebo; Test type: Superiority or Other; p = 0.0204, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted percent difference for saxagliptin 5 mg vs placebo in Week 12 (LOCF) to baseline ratio. Adjusted for baseline; Adjusted Percent Difference = 27.9, 95% CI 2-sided [4.2 to 57.1] — ANCOVA model: logarithm(post/pre) = logarithm(pre) treatment

3. Other Pre Specified Outcome: Overall Summary of Adverse Events (AEs) Serious AEs (SAEs), Discontinuations, and Deaths During the ST + LT Treatment Period
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event. Related events=relationship of certain, probable, possible, or missing.
Time Frame: 116 weeks
Population: Treated participants
Measure: Number; unit: participants
Arm/Group | Saxagliptin 5 mg | Placebo / Metformin
Number analyzed (Participants) | 20 | 16
participants
  At Least 1 AE | 17 | 14
  At Least 1 Related AE | 7 | 6
  Deaths | 0 | 0
  At Least 1 SAE | 1 | 2
  At Least 1 Related SAE | 0 | 0
  Discontinuations Due to SAEs | 0 | 1
  Discontinuations Due to AEs | 0 | 2

4. Other Pre Specified Outcome: Marked Laboratory Abnormalities - During ST + LT Treatment Period
Description: A laboratory value was considered a marked abnormality if it is outside the pre-defined criteria for marked abnormality and the on-treatment value was more extreme (farther from the limit) than the baseline value. Pre-Rx=pretreatment; ULN=upper limit of normal; ALP=alkaline phosphatase; AST=aspartate aminotransferase; ALT=alanine aminotransferase; BUN=blood urea nitrogen; unspec.=unspecified; sodium serum low: <0.9 x Pre-Rx & <=130mEq/L / high: >1.1 x Pre-Rx & >=150mEq/L; potassium, serum low: <=0.8 x Pre-Rx & >=6.0mEq/L / high: 1.2 x Pre-Rx & >=6.0mEq/L; LLN=lower limit of normal.
Time Frame: 116 weeks
Population: Number of Participants Analyzed=Treated participants; n=number of treated subjects with baseline value and at least one value during the ST + LT treatment period.
Measure: Number; unit: participants
Arm/Group | Saxagliptin 5 mg | Placebo / Metformin
Number analyzed (Participants) | 20 | 16
participants
  Hemoglobin < 8 g/dL (n=0, 0) | 0 | 0
  Hematocrit < 0.75 x pre-Rx (n=0, 0) | 0 | 0
  Platelets < 50 x 10^9 c/L (n=0, 0) | 0 | 0
  Platelets > 1.5 x ULN (n=0, 0) | 0 | 0
  Leukocytes < 2 x 1000 c/uL (n=0, 0) | 0 | 0
  Neutrophils+Bands <1x1000 c/uL (n=18, 0) | 1 | 0
  Eosinophils >0.9x1000 c/uL (n=18, 0) | 1 | 0
  Lymphocytes <=0.75x1000 c/uL (n=18, 0) | 2 | 0
  ALP >3 x pre-Rx and >ULN (n=0, 0) | 0 | 0
  AST >3 x ULN (n=0, 0) | 0 | 0
  AST >5 x ULN (n=0, 0) | 0 | 0
  ALT >3 x ULN (n=0, 0) | 0 | 0
  ALT >5 x ULN (n=0, 0) | 0 | 0
  Bilirubin Total >2mg/dL (n=0, 0) | 0 | 0
  BUN >2 x pre-Rx and >ULN (n=0, 0) | 0 | 0
  Creatinine >2.5 mg/dL (n=0, 0) | 0 | 0
  Glucose, Serum Fasting < 50 mg/dL (n=0, 0) | 0 | 0
  Glucose, Serum Fasting > 500 mg/dL (n=0, 0) | 0 | 0
  Glucose, Serum Unspec. < 50 mg/dL (n=0, 0) | 0 | 0
  Glucose, Serum Unspec. > 500 mg/dL (n=0, 0) | 0 | 0
  Glucose, Plasma Fasting <50 mg/dL (n=0, 0) | 0 | 0
  Glucose,Plasma Fasting >500 mg/dL (n=0, 0) | 0 | 0
  Glucose, Plasma Unspec. <50 mg/dL (n=0, 0) | 0 | 0
  Glucose, Plasma Unspec. >500 mg/dL (n=18, 16) | 8 | 9
  Sodium, Serum Low (see description) (n=0, 0) | 0 | 0
  Sodium, Serum High (see description) (n=0, 0) | 0 | 0
  Potassium, Serum Low (see description) (n=0, 0) | 0 | 0
  Potassium, Serum High (see description) (n=0, 0) | 0 | 0
  Chloride < 90 mEq/L (n=0, 0) | 0 | 0
  Chloride > 120 mEq/L (n=0, 0) | 0 | 0
  Albumin < 0.9 LLN (n=0, 0) | 0 | 0
  Creatine Kinase > 5 x ULN (n=18, 16) | 1 | 1
  Uric Acid > 1.5 x ULN (n=0, 0) | 0 | 0
  Protein Urine, >=2-4 (n=0, 0) | 0 | 0
  Blood Urine >=2-4 (n=18, 0) | 1 | 0
  Red Blood Cells Urine >=2-4 (n=0, 0) | 0 | 0
  White Blood Cells Urine >=2-4 (n=0, 0) | 2 | 1

ADVERSE EVENTS:
Time Frame: Short term period (up to 12 weeks) + long term period (up to 104 weeks)
Groups:
- PLACEBO/METFORMIN: Placebo Tablet, Oral, 0 mg, once daily, up to 12 weeks (short term); Metformin Tablet, Oral, 500 mg titrated to 1000 mg, once daily, up to 104 weeks (long term)
- SAXAGLIPTIN 5 MG: Tablet, Oral, 5 mg, once daily, up to 12 weeks (short term); Tablet, Oral, 5 mg, once daily, up to 104 weeks (long term)
Arm/Group | PLACEBO/METFORMIN | SAXAGLIPTIN 5 MG
Serious Adverse Events (participants affected / at risk) | 2/16 | 1/20
Other Adverse Events (participants affected / at risk) | 14/16 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PLACEBO/METFORMIN (N=16) | SAXAGLIPTIN 5 MG (N=20)
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
CHEST DISCOMFORT (General disorders) | 0 | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PLACEBO/METFORMIN (N=16) | SAXAGLIPTIN 5 MG (N=20)
EYE IRRITATION (Eye disorders) | 1 | 0
LACRIMATION INCREASED (Eye disorders) | 0 | 1
CARDIAC MURMUR (Investigations) | 0 | 1
URINE OUTPUT DECREASED (Investigations) | 0 | 1
BLOOD PRESSURE INCREASED (Investigations) | 1 | 0
EOSINOPHIL COUNT INCREASED (Investigations) | 0 | 1
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 1
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0
HAEMATOMA (Vascular disorders) | 1 | 0
HOT FLUSH (Vascular disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 2 | 0
PERIPHERAL COLDNESS (Vascular disorders) | 1 | 0
STRESS (Psychiatric disorders) | 0 | 1
INSOMNIA (Psychiatric disorders) | 1 | 0
AGITATION (Psychiatric disorders) | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 1 | 0
SEASONAL ALLERGY (Immune system disorders) | 1 | 0
TREMOR (Nervous system disorders) | 0 | 1
AGEUSIA (Nervous system disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 3 | 5
DIZZINESS (Nervous system disorders) | 1 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 1
PRESYNCOPE (Nervous system disorders) | 1 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 2
HYPOAESTHESIA (Nervous system disorders) | 1 | 1
SINUS HEADACHE (Nervous system disorders) | 1 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 3 | 2
VOMITING (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 2
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 2
FLATULENCE (Gastrointestinal disorders) | 2 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 0
FAECES DISCOLOURED (Gastrointestinal disorders) | 0 | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 2 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 0 | 1
MIDDLE EAR EFFUSION (Ear and labyrinth disorders) | 0 | 1
CYSTITIS (Infections and infestations) | 0 | 1
RHINITIS (Infections and infestations) | 0 | 1
INFLUENZA (Infections and infestations) | 5 | 0
SINUSITIS (Infections and infestations) | 0 | 3
BRONCHITIS (Infections and infestations) | 1 | 0
BACTERIURIA (Infections and infestations) | 0 | 1
INFECTED CYST (Infections and infestations) | 1 | 0
LABYRINTHITIS (Infections and infestations) | 0 | 1
TOOTH ABSCESS (Infections and infestations) | 1 | 0
OTITIS EXTERNA (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 2
NASOPHARYNGITIS (Infections and infestations) | 3 | 3
KIDNEY INFECTION (Infections and infestations) | 1 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 1
HELICOBACTER INFECTION (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 3
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
BLADDER DILATATION (Renal and urinary disorders) | 0 | 1
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 0 | 2
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN LESION (Skin and subcutaneous tissue disorders) | 2 | 0
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 1
PROSTATITIS (Reproductive system and breast disorders) | 1 | 0
GYNAECOMASTIA (Reproductive system and breast disorders) | 0 | 1
TESTICULAR PAIN (Reproductive system and breast disorders) | 0 | 1
UTERINE PROLAPSE (Reproductive system and breast disorders) | 0 | 1
ENDOMETRIAL HYPERTROPHY (Reproductive system and breast disorders) | 1 | 0
PROSTATIC CALCIFICATION (Reproductive system and breast disorders) | 0 | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
HEAT EXHAUSTION (Injury, poisoning and procedural complications) | 0 | 1
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 1
POST PROCEDURAL SWELLING (Injury, poisoning and procedural complications) | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 2
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 5
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 2
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 1
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PAIN (General disorders) | 1 | 0
FATIGUE (General disorders) | 2 | 2
CHEST PAIN (General disorders) | 1 | 0
HERNIA PAIN (General disorders) | 0 | 1
CHEST DISCOMFORT (General disorders) | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 2
INFUSION SITE PAIN (General disorders) | 2 | 4
INFUSION SITE DISCOMFORT (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.